CLINICAL TRIAL: NCT04712084
Title: Postoperative Atelectasis Prevention by Application of PEEP and Pressure Support Ventilation: a Prospective Randomized Controlled Trial
Brief Title: Postoperative Lung Collapse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lennart Magnusson (Other)
Responsible Party: Sponsor-Investigator, Lennart Magnusson, MD Lennart Magnusson PhD, PD, Hôpital Fribourgeois
Organization: Hôpital Fribourgeois (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: anesth2020
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Atelectasis
Keywords: anesthesia, general
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: prospective double-blinded study Randomization was performed when spontaneous ventilation resumed at the end of the surgery
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient during general anesthesia are not aware of the technique applied. The radiologist calculating the surface of atelectasis is not aware of the technique applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Extubation procedure following standard of care
- Pressure support group (Experimental): Extubation procedure is performed with 100% of O2 but with application of positive pressure before and after extubation
  Interventions: Procedure: Positive pressure

INTERVENTIONS:
Procedure: Positive pressure — Inspiratory support of 8 cmH2O was applied associated with PEEP at 6 cmH2O. After extubation, same support was applied by facemask for 3 minutes
  Arms: Pressure support group

SUMMARY:
General anaesthesia is known to promote lung collapse (atelectasis) which will persist in the postoperative period. Inflating the lung to a pressure of 40 cmH2O, called a vital capacity manoeuvre (VCM), performed a few minutes before extubation followed by the use of 40% of O2 will prevent postoperative atelectasis formation. This is not the case if VCM is followed by application of 100% of O2. However the use of 100% of O2 before tracheal extubation is still recommended for safety reason. Application of PEEP associated with pressure controlled ventilation before intubation prevents atelectasis formation despite the use of 100% of O2. The goal of our study was to show that performing a VCM 15 minutes before arousal followed by application of PEEP and pressure support ventilation (PSV) before and after tracheal extubation will prevent the recurrence of atelectasis despite the use of 100% of O2.

Materials and Methods With the ethic committee for research on human beings approval, the investigators randomly assigned 16 non-obese patients scheduled for a gynaecological laparoscopic surgery in two groups. At the end of the surgery the investigators performed a VCM (40cmH2O applied for 12 seconds), then O2 was increased to 100% in both groups. In the patients of the study group, a PEEP of 6 cmH2O was applied associated with a PSV of 8 cmH2O. This was continued after the extubation for 3 minutes. The O2 was then decreased to 40% and, when the expired oxygen saturation was < 50%, PEEP and PSV were removed. For the patients in the control group, no positive pressure was applied during spontaneous ventilation (PEEP = 0 and no PSV). The atelectasis were then measured by computed tomographic scanning.

DETAILED DESCRIPTION:
This is a prospective double-blinded study with prior informed written consent obtained from all patients.

Study Population Patients aged 18 to 65 years, American Society of Anesthesiologist (ASA) physical status classification I to III, undergoing gynaecological laparoscopic surgery under general anaesthesia were included in this prospective, randomised, double-blinded study.

Exclusion criteria were severe pulmonary disease, body mass index (BMI) more than 30 kg /m2 or less than 17, pregnancy or any other disease for which hypoxemia could be harmful. If the delay between extubation and the computed tomography (CT) scan was over 20 minutes, patients were also excluded.

Study treatments No premedication was given. General anaesthesia was standardized for all patients. Standard monitoring was applied. General anaesthesia was induced intravenously with fentanyl 1 to 2 μg/kg, propofol 2 to 3 mg/kg, and rocuronium 0.6 mg/kg. The airways were secured by endotracheal intubation.

Desflurane was used for maintenance at 1 minimal alveolar concentration (MAC) in 40% oxygen and air. Additional rocuronium was injected in order to maintain a train-of-four ratio (TOF ratio) between 0 and 1/4. Supplemental fentanyl was administered in order to maintain blood pressure and/or heart rate values within a range of 20% compared to baseline values.

For ventilation, the investigators used pressure controlled mode with tidal volume guaranteed (pressure controlled - guaranteed volume, General Electrics Datex-Ohmeda Aisys®). The settings of ventilation were, tidal volume 6-8 ml/kg (ideal body weight), frequency 10 - 20 per min. (expired CO2 5.3 - 5.8 kPa), PEEP of 6 cmH2O and I:E ratio 1:2.

Fifteen minutes before the end of the surgery, a VCM (40cmH2O applied for 12 seconds) was performed, then O2 was increased to 100% in both groups. Sugamadex (4 mg/kg if TOF <2/4, 2 mg/kg if TOF >2/4) was administered in order to reverse neuromuscular block. General anaesthesia was continued until TOF ratio > 90%.

Randomization was performed when spontaneous ventilation resumed. In the study group, inspiratory support of 8 cmH2O was applied associated with PEEP at 6 cmH2O. After extubation, same support was applied by facemask for 3 minutes. O2 was then decreased to 40% and, when the expired oxygen fraction was < 50%, PEEP and PSV were switched off.

In the control group, no positive pressure and no PEEP were applied during spontaneous ventilation and 100% of O2 was applied for 3 minutes after extubation with a facemask.

Patients were then transported to the CT scan breathing 40% of O2 via a facemask. The peripheral oxygen saturation was continuously monitored by pulse oximetry. Postoperative pain management consisted of the residual effect of intraoperative fentanyl and paracetamol if required.

Measurements Whole lung CT scan with a special low doses protocol was obtained at end-expiratory position (at functional residual capacity).

Measurement was performed for all the lung and the lungs were also divided in 3 zones (upper, middle and lower). Each right and left lung surfaces were extracted and a window setting of -1000 to +100 Hounsfield Units (HU) was selected to assess the total lung surface. A threshold of -1000 to -500 HU was applied to quantify the amount of normally ventilated lung, a second threshold of -500 to -100 HU was chosen to establish the surface of poorly ventilated lung, and a third threshold of -100 to +100 HU was set to measure the surface of atelectatic lung area. The right and left lungs surface were summed and reported to the total lung surface(18).

Study Outcome The primary outcome was diminution of atelectatic and poorly ventilated lung volume in the study group compared to the control group.

Statistical Analysis Values are expressed as mean +/- SD. Baseline results and atelectatic surface were compared by a one-way analysis of variance for continuous variables and with X2 for discrete variables. P < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patient undergoing gynaecological laparoscopic surgery under general anesthesia

Exclusion Criteria:

* BMI > 30 kg/m2 or < 17 kg/m2
* pregnancy; hypoxemic disease
* Delay between extubation and CT-scan > 20 minutes

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2014-07-22 (Actual); Study Completion 2014-07-22 (Actual)

PRIMARY OUTCOMES:
Atelectatic surface | 10 - 20 minutes after extubation
  Whole lung CT scan with a special low doses protocol was obtained at end-expiratory position (at functional residual capacity)

CONTACTS AND LOCATIONS:
Overall Officials: Lennart Magnusson, Study Director — Hopital cantonal Fribourg

IPD SHARING:
Plan to Share IPD: No